CLINICAL TRIAL: NCT01129609
Title: Talent Converter Post-Approval Study
Status: Terminated | Type: Observational
Why Stopped: Low subject enrollment due to obseleted product.
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: Investigational Plan #119
Record Dates: First submitted 2010-04-29; First posted 2010-05-24 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Post-approval observation of patients being treated according to the indications for use for the Talent Converter Stent Graft
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Successful Secondary Endovascular Treatment
  Interventions: Device: Talent Converter Stent Graft and Talent Occluder with Occluder Delivery System

INTERVENTIONS:
Device: Talent Converter Stent Graft and Talent Occluder with Occluder Delivery System — All subject enrolled will be attempted to be treated with or will be treated with the Talent Converter Stent Graft

SUMMARY:
The primary endpoint is successful secondary endovascular treatment with the Talent Converter stent graft of subjects having received prior endovascular repair of infrarenal abdominal aortic or aortoiliac aneurysms using the Talent or AneuRx Bifurcated Stent Grafts, in which there is inadequate proximal fixation, seal, overlapping of modular components or unattainable contralateral limb cannulation.

Treatment success is defined as a composite of successful vessel access, successful insertion of the delivery system, successful deployment of the Converter stent graft at the intended treatment site and absence of Type I endoleak at the 1 month follow-up visit.

DETAILED DESCRIPTION:
Converter PAS is an observational study. Patients will receive treatment regardless of study participation. In some cases, patients will be enrolled retrospectively, post implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects in whom a vessel access procedure was/will be performed with the attempted introduction of the Talent Converter Stent Graft for use according to the indications for use in the Instructions for Use (IFU) 0-365 days prior to enrollment.
2. Subjects who are able to understand the nature of the study and give voluntary informed consent.
3. Subjects who are available for follow-up visits.
4. Subjects 18 years of age or older.

Exclusion Criteria:

1. Subjects in whom an attempted treatment was/will be performed with the Talent Converter Stent Graft other than (i.e., primary AUI) as a secondary endovascular intervention for patients having received prior endovascular repair with either a Talent or AneuRx bifurcated stent graft.
2. Subjects in whom an attempted treatment was/will be performed with the Talent Converter Stent Graft as a secondary endovascular intervention for patients having received prior endovascular repair with a bifurcated stent graft other than (i.e., Cook Zenith or Gore Excluder) a Talent or AneuRx bifurcated stent graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who are treated with the Talent Converter Stent Graft according to the indications for use
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2013-06 (Actual); Study Completion 2017-09-29 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Subjects: Talent Converter Stent Graft and Talent Occluder with Occluder Delivery System: All subject enrolled will be attempted to be treated with or will be treated with the Talent Converter Stent Graft
Period: Overall Study
Arm/Group | All Enrolled Subjects
Started | 20
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: All Enrolled Subjects
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Successful Secondary Endovascular Treatment
Description: The outcome measure is successful secondary endovascular treatment with the Talent Converter stent graft where treatment success is defined as successful vessel access, successful insertion of the delivery system, successful deployment of the Converter stent graft at the intended treatment site and absence of Type I endoleak at the 1 month follow-up visit.
Time Frame: 30 days
Population: Number of Participants with Successful Secondary Endovascular Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 20
Participants | 17

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- All Enrolled Subjects: Talent Converter Stent Graft and Talent Occluder with Occluder Delivery System: All Subjects enrolled will be attempted to be treated with or will be treated with the Talent Converter Stent Graft.
Arm/Group | All Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 10/20
Serious Adverse Events (participants affected / at risk) | 11/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Device Dislocation (General disorders) | 1 (1)
Stent-Graft Endoleak (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Failure To Thrive (Metabolism and nutrition disorders) | 1 (1)
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Parkinson's Disease (Nervous system disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1)
Nephropathy Toxic (Renal and urinary disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aneurysm Ruptured (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
FDA allowed for early termination of the Talent Converter PAS because the device is no longer being manufactured, and exsisting inventory of the device has since expired, thus no statistical conclusions will be derived due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No